CLINICAL TRIAL: NCT07372508
Title: GALACTIC 1 - Glasgow Low-dose CT and AI-based Diagnostics to Case Find Lung Cancer and Other Cardio-respiratory Long-term Conditions - Feasibility Study
Brief Title: Glasgow Low-dose CT and AI-based Diagnostics to Case Find Lung Cancer and Other Cardio-respiratory Long-term Conditions - Feasibility Study
Acronym: GALACTIC-1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INGN25HS173; IRAS: 357735 (Other: IRAS)
Record Dates: First submitted 2026-01-09; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): All patients
  Interventions: Diagnostic Test: Low dose Chest CT

INTERVENTIONS:
Diagnostic Test: Low dose Chest CT — Low dose Chest CT

SUMMARY:
Lung cancer is one of the most common and serious cancers in Scotland and is often diagnosed at a late stage. Early detection is crucial to improving survival rates. The value of screening for lung cancer with low-dose CT (LDCT) scans has been established, and these scans can also identify other diagnoses earlier.

Additional tests undertaken alongside the CT scan may add value to the lung cancer screening program being rolled out. This study aims to explore the feasibility and utility of a lung cancer screening program with added heart and breathing tests within a single clinic visit.

A Lung Health Check will be offered to people at higher risk of lung cancer, specifically those aged 55-74 with a history of cigarette smoking. This will include a quick and painless LDCT scan, which uses a small amount of radiation to create detailed images of the lungs to detect lung cancer at an early and more treatable stage.

In this "GALACTIC-1" study, the investigators will explore whether structured reporting of the CT scan, combined with additional tests (blood sample, ECG heart trace, and spirometry breathing test), can help identify conditions such as chronic obstructive pulmonary disease (COPD), lung scarring (pulmonary fibrosis), coronary artery disease, heart failure, and early signs of bone fractures (osteoporosis). This enhanced Lung Health Check may improve overall health by identifying and allowing early management of these conditions.

The investigators plan to use the data from the "GALACTIC-1" study to explore AI performance by comparing it to reporting done by doctors. The results will help shape future rollout of lung cancer screening across Scotland, ensuring it is effective, efficient, and beneficial.

The investigators will also have a focus group with patients and interviews with NHS staff to understand their opinions on the screening.

ELIGIBILITY:
Inclusion Criteria:

* Resident in South Sector NHS GG&C.
* Capacity to undertake informed consent.
* No active cancer other than non-melanoma skin cancer, monitored localised prostate cancer or localised treated breast cancer.
* Aged 55-74 at date of invitation.
* Smoking history: current tobacco smoker or ex-smoker with >20 pack year history and <15 years from quit date.

Exclusion Criteria:

* CT thorax scan undertaken in prior 12 months.
* Does not have capacity to give consent (standard criteria for assessing capacity apply).
* Aged <55 or >74 years of age at date of invitation
* Weight exceeds restrictions for scanner (>200kg).
* Unable to lie flat.
* People who are pregnant.
* Active symptoms of possible lung cancer

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-09-02 (Estimated); Study Completion 2028-09-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible invited participants who receive all components of the combined low-dose CT (LDCT) screening and AI-assisted cardiorespiratory diagnostic tests within the study active period. | 6 months
  Number of patients successfully screened per protocol within recruitment timelines

SECONDARY OUTCOMES:
Sensitivity of LDCT for detecting confirmed lung cancer (proportion of patients with lung cancer correctly identified as positive). | Baseline
Specificity of LDCT for detecting confirmed lung cancer (proportion of patients without lung cancer correctly identified as negative). | Baseline
Lung cancer detection rate | Baseline
  Proportion of participants found to have lung cancer
Stage distribution of detected lung cancers | Baseline
  The proportion detected at Stage I/II vs. Stage III/IV
Detection rate of undiagnosed COPD and/or emphysema in participants. | Baseline
Detection rate of undiagnosed interstitial lung abnormalities (ILA) and pulmonary fibrosis in participants. | Baseline
Detection rate of undiagnosed significant coronary artery disease (CAD) in participants | Baseline
Detection rate of undiagnosed heart failure - radiological, ECG or biomarker (elevated NT-proBNP) indicators requiring further evaluation in participants. | Baseline
Detection rate of undiagnosed osteoporotic fractures in participants. | Baseline
Impact of addressable long-term condition case-finding on subsequent investigations, preventative therapy initiation and clinical outcomes. | Year 1 and Year 2
  Accessible health records, investigation requests, prescriptions, hospital admissions and survival at year 1 and year 2 post Galactic-1 clinic will be reviewed to determine the impact the LDCT had on the patient's care.
Performance and potential utility of AI-based radiology co-reporting of lung cancer screening CT scans | Baseline
  Number of radiology reports which agree with the AI report
Acceptability and qualitative evaluation | Baseline
  Participant experience questionnaires will be collected during GALACTIC-1 clinic to provide an overview of experienced acceptability at the time of clinic attendance. Additional focus group or semi-structured interviews will be conducted.
The potential cost-effectiveness of AI-detection of early-stage lung cancer as well as other conditions such as COPD, pulmonary fibrosis, coronary artery disease, heart failure, and osteoporotic fractures | Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Chris Carlin, Principal Investigator — NHSGGC
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided